CLINICAL TRIAL: NCT06283589
Title: The SEAPORT 1 Study: An Open-label Exploratory Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of INZ-701 in Study Participants With End-Stage Kidney Disease Undergoing Hemodialysis
Brief Title: The SEAPORT 1 Study: Evaluation of the Safety and Tolerability of INZ-701 in Adults With End-Stage Kidney Disease Undergoing Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inozyme Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INZ701-401
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Calciphylaxis
Keywords: calcific uremic arteriolopathy; calcinosis cutis; calcification; calcium metabolism disorders; mineral bone disorder (MBD); fusion protein; vascular calcification; end stage renal disease (ESKD); chronic kidney disease (CKD); calcinosis
MeSH Terms: conditions — Calciphylaxis; Calcinosis Cutis; Calcinosis; Calcium Metabolism Disorders; Vascular Calcification; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The SEAPORT 1 (INZ701-401) study is a Phase 1, open-label, multi-center study to evaluate the safety, pharmacokinetics, and pharmacodynamics of multiple doses of INZ-701, given once per week over 4 weeks, in study participants with end-stage kidney disease undergoing hemodialysis.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INZ-701 (Experimental): The study consists of a 26-day treatment period where the dose of INZ-701 will be 1.8 mg/kg once weekly. INZ-701 will be administered as a subcutaneous injection once weekly for 4 weeks on Days 3, 10, 17, and 24. The study participant's post-hemodialysis body weight on Day 1 will be used to calculate the dose to be administered.
  Interventions: Drug: INZ-701

INTERVENTIONS:
Drug: INZ-701 — Recombinant fusion protein that contains the extracellular domains of human ENPP1 coupled with an Fc fragment from an immunoglobulin gamma-1 (IgG1) antibody.
  Other Names: (rhENPP1-Fc).

SUMMARY:
The purpose of this study is to determine if multiple doses of INZ-701, given once per week over 4 weeks are safe and increase pyrophosphate (PPi) levels in hemodialysis-dependent (HD) end stage kidney disease (ESKD) study participants who have low PPi levels. In addition, the effect of hemodialysis on the pharmacokinetics of INZ-701 and PPi levels will be evaluated.

DETAILED DESCRIPTION:
INZ-701 is an ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) recombinant fusion protein in development for the treatment of calciphylaxis. The SEAPORT 1 (INZ701-401) Study is a Phase 1, open-label study to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple doses of INZ-701 in study participants aged >18 to < 70 years with HD-dependent ESKD. Anticipated enrollment in the study is up to 10 study participants. The purpose of this study is to determine if INZ-701 increases PPi levels, as well as assess the PK/ PD characteristics of INZ-701 in patients with clinically low PPi levels.

The study will consist of a Screening Period lasting up to 30 days, a Treatment and Assessment Period lasting 26 days, an End of Study (EOS) Visit 30- or 60- days after the last dose of INZ-701, , and a Follow-Up Period lasting up to 365 days after the last dose During the Follow-Up Period, safety, PPi, ENPP1 activity, anti-drug antibodies (ADA) assessments, and genetic testing will be conducted. Participants may be followed for > 1 year if they have increasing ADA titers or have serious adverse events (SAEs) related to ADAs as determined by the Sponsor

ELIGIBILITY:
Inclusion Criteria:

Individuals meeting the following inclusion criteria may participate:

1. Study participants must provide written or electronic consent after the nature of the study has been explained, and prior to any research-related procedures, per International Council for Harmonisation (ICH) Good Clinical Practice (GCP)
2. Have ESKD and are receiving HD treatment
3. Are compliant with receiving 3 treatments of HD per week with a functioning arteriovenous (AV) fistula, AV graft, or central venous catheter
4. PPi level <700 nmol/L at Screening
5. Must be willing and able to comply with the diet prescribed by their treating physician and/or the Investigator
6. Male or female aged >18 years to <70 years
7. Women of child-bearing potential (WOCBP) as defined in Clinical Trials Coordination Group (CTFG 2020) and provided in Appendix B, must have a negative serum pregnancy test at Screening and within 3 days of INZ-701 administration
8. WOCBP and partners of fertile males who are WOCBP must be using or agree to use one highly effective form of contraception (per CTFG 2020) and a barrier method from at least 1 month before the first dose of INZ-701 to 30 days after the last dose (greater than 5 half-lives of INZ-701). WOCBP and partners of fertile males who are WOCBP must also agree to not donate ova from the time of the first INZ-701 dose to 30 days after the last dose.
9. Males who are sexually active must agree to use condoms from the time of the first INZ-701 dose to 30 days after the last dose. Males must also agree to not donate sperm from the time of the first INZ-701 dose to 30 days after the last dose.
10. In the opinion of the Investigator, study participants are able and willing to complete all study procedures per protocol.

Exclusion Criteria:

Individuals meeting any of the following exclusion criteria may not participate:

1. Study participants receiving other types of dialysis than HD (eg, peritoneal dialysis, hemodiafiltration)
2. Study participants who are hospitalized
3. In the opinion of the Investigator, presence of any clinically significant disease or laboratory abnormality that may impact study participation and/or confound interpretation of the study results
4. Malignancy within the last year, except non-melanoma skin cancers or cervical carcinoma in situ
5. Advanced liver disease manifesting as liver cirrhosis
6. Myocardial infarction, stroke, or congestive heart failure requiring hospitalization within the last 6 months
7. Known intolerance to INZ-701 or any of its excipients
8. Weight >125 kg
9. Concurrent participation in another interventional clinical study and/or receipt of any other investigational new drug within 5 half-lives of the last dose of the other investigational product or from 4 weeks prior to the first dose of INZ-701, whichever is longer, or use of an investigational device, through completion of participation in the study

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Determine if INZ-701 increases PPi levels | 26 days (Treatment Period)
  For each participant, plasma PPi will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time to determine if there's been a change.

SECONDARY OUTCOMES:
Assess the Time to Maximum Serum Concentration (Tmax) | 26 days (Treatment Period)
  For each participant, the maximum concentration of INZ-701 in the serum will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.
Assess the Maximum Serum Concentration (Cmax) of INZ-701 | 26 days (Treatment Period)
  For each participant, the maximum concentration of INZ-701 in the serum will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.
Assess the Area under the concentration-time curve over the dosing interval (AUCtau) | 26 days (Treatment Period)
  For each participant, variation of concentration of INZ-701 in the serum will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.
Assess the Clearance after extravascular administration of drug (CL/F) | 26 days (Treatment Period)
  For each participant, clearance of INZ-701 from the body will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.
Assess ENPP1 Activity | 26 days (Treatment Period)
  For each participant, ENPP1 activity is a measurement of INZ-701 activity in human serum using a chromogenic based method.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — Inozyme Pharma
Locations (2):
- United States (2):
  - South Florida Nephrology Research, Coral Springs, Florida
  - Elixia Health, Hollywood, Florida